CLINICAL TRIAL: NCT06715579
Title: Cardiac Angiosarcoma International Registry
Acronym: CAIR
Status: Not yet recruiting | Type: Observational
Sponsor: Immune Oncology Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMMONC0020
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Angiosarcoma
Keywords: Cardiac Angiosarcoma; Angiosarcoma; Hemangiosarcoma; Epithelioid Hemangiosarcoma; Primary Cardiac Sarcoma
MeSH Terms: conditions — Hemangiosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Primary cardiac angiosarcomas (PCA) are highly aggressive malignant heart tumors arising from the endothelial cells (ECs) lining the blood vessels of the heart and account for approximately 25%-30% of all primary cardiac malignancies. It is considered to be the most fatal and aggressive primary cardiac malignancy. This international registry aims to establish a large multicenter database of patients with cardiac angiosarcoma. Our objectives are:

1. Collect clinical data, including demographics, medical history, treatments, and outcomes, to build a comprehensive database.
2. Analyze data to evaluate and identify genetic, environmental, or lifestyle risk factors for cardiac angiosarcoma.
3. Evaluate the effectiveness of various treatments (surgery, chemotherapy, immunotherapy, radiation) to inform best practices.
4. Develop evidence-based guidelines and recommendations for prevention, diagnosis, treatment, and management based on registry data.

DETAILED DESCRIPTION:
Primary cardiac angiosarcoma arises directly within the heart, unlike secondary cardiac tumors that originate from elsewhere in the body. While it predominantly affects the right side of the heart, particularly the right atrium, it can also impact other cardiac chambers and structures. The characteristic feature of cardiac angiosarcoma is the rapid formation of abnormal blood vessels that invade the myocardium, leading to the destruction of healthy heart tissue.The five-year survival rate for patients with primary cardiac angiosarcoma (PCA) is reported to be around 14%. In contrast, familial variants of this malignancy exhibit even more severe outcomes, with a mean survival rate of only 4 months.

Establishing an international registry for cardiac angiosarcomas is crucial for several reasons:

* The registry will facilitate a comprehensive understanding of the clinical characteristics, treatment responses, and outcomes associated with cardiac angiosarcoma. By collecting data from diverse populations, researchers can identify patterns and factors that influence survival rates. It is crucial to better understand the growth rates and risk factors associated with cardiac angiosarcoma and to make the disease more manageable.
* The international registry will enable the latest advancements in oncology and related medical fields to be incorporated into clinical practice. It will provide a platform for developing and conducting clinical trials aimed at improving treatment strategies and increasing survival rates for patients with cardiac angiosarcoma.
* Finally, with data from various institutions and countries, the registry will promote collaboration among healthcare professionals, researchers, and institutions dedicated to improving outcomes for patients with this rare malignancy.

Creating an international registry for cardiac angiosarcoma is crucial for better understanding this aggressive cancer. It will help address the rising cancer burden and support research and treatment advancements that could improve patient survival rates and prevention.

The following data will be collected through questionnaires:

1. Patient characteristics
2. Characteristics of Primary Cardiac Angiosarcomas
3. Details of the diagnosis and treatment
4. Complications and late effects of treatment
5. Outcomes and follow-up information

Quality control and data management will be done by the Immune Oncology Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Histological Confirmation: A confirmed diagnosis of cardiac angiosarcoma through histopathological examination, including subtypes such as hemangiosarcoma and epithelioid hemangiosarcoma.
* Diagnosis Timing: Eligible patients must have been diagnosed between January 2015 and January 2035.
* Geographical Representation: Participants should be from diverse geographical locations to ensure a comprehensive understanding of the disease across different populations.
* Treatment Status: Patients who have received any treatment (surgery, chemotherapy, immunotherapy or radiation) for cardiac angiosarcoma may be included to evaluate treatment outcomes.
* Informed Consent: For prospective patients, informed consent must be obtained before they are included in the registry.
* Clinical Data Availability: Relevant clinical data, including demographics, tumor characteristics (size, location), treatment regimens, and outcomes, must be available for analysis.
* Follow-Up Willingness: Participants should be willing to undergo follow-up assessments as part of the registry's data collection efforts.

Exclusion Criteria:

* Patients who decline to provide informed consent.
* Cases where cardiac involvement is secondary to another primary malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with Cardiac Angiosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2035-05 (Estimated); Study Completion 2035-05 (Estimated)

PRIMARY OUTCOMES:
6-month overall survival | 6 months

SECONDARY OUTCOMES:
1-year overall survival | 1 year
6-month progression free survival | 6 months
1-year progression free survival | 1 year
3-year progression free survival | 3 years
6-month event-free survival | 6 months
1-year event-free survival | 1 year
3-year event-free survival | 3 years
Complete remission rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shushan Hovsepyan, MD, Principal Investigator — Immune Oncology Research Institute, Yerevan, Armenia; Amalya Sargsyan, MD, Study Chair — Immune Oncology Research Institute, Yerevan, Armenia; Ruzanna Papyan, MD, Study Director — Immune Oncology Research Institute, Yerevan, Armenia
Locations (1):
- Yeolyan Hematology and Oncology Center, Yerevan, Armenia